CLINICAL TRIAL: NCT07348757
Title: Comparison of rFSH Alone Versus rFSH+rLH in Dydrogesterone-Based Progestin Protocol Cycles
Brief Title: rFSH vs rFSH+rLH in Dydrogesterone-Based Progestin Protocol: A Prospective Study
Acronym: DYG-GONA
Status: Recruiting | Type: Observational
Sponsor: Centrum Clinic IVF Center (Other)
Responsible Party: Principal Investigator, Emre Göksan Pabuçcu, Prof. Dr., Centrum Clinic IVF Center
Other Study IDs: 2025-11
Record Dates: First submitted 2025-11-19; First posted 2026-01-16 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: InVitro Fertilization; Gonadotropins
Keywords: gonadotropins; invitro fertilization; pregnancy; ppos

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recombinant FSH Only Group: Recombinant FSH (rFSH) Group - Additional Information
  Participants in this cohort will undergo ovarian stimulation using recombinant follicle-stimulating hormone (rFSH) alone, following routine IVF clinical practice. Dydrogesterone will be initiated on Cycle Day 2 as part of the standard PPOS (Progestin-Primed Ovarian Stimulation) protocol to prevent premature LH surge. Follicular development will be monitored with ultrasound and serum hormone levels, and the timing of final oocyte maturation and oocyte pick-up will follow standard clinical procedures. No additional medications or interventions will be administered beyond those routinely used for IVF treatment.
- Recombinant FSH Plus Recombinant LH Group: Recombinant FSH Plus Recombinant LH (2:1 Combination) Group - Additional Information
  Participants in this cohort will receive a combination of recombinant follicle-stimulating hormone (rFSH) and recombinant luteinizing hormone (rLH) in a fixed 2:1 ratio, as routinely used in clinical IVF practice. Dydrogesterone will be initiated on Cycle Day 2 according to the standard PPOS (Progestin-Primed Ovarian Stimulation) protocol to prevent premature LH surge. Follicular development will be monitored through ultrasound examinations and serum hormone measurements, and final oocyte maturation and oocyte retrieval will be performed following standard clinical procedures. No additional treatments or study-specific interventions will be administered beyond those normally used in IVF care.

SUMMARY:
This study aims to compare two commonly used hormone treatments for women undergoing IVF. All participants will receive a stimulation protocol that includes dydrogesterone, a medication used to safely control natural hormone surges during treatment. The study will observe women who are treated either with recombinant FSH alone or with a combination of recombinant FSH and recombinant LH-both routinely used options in our clinic.

Investigators will prospectively monitor how these treatments affect the growth of ovarian follicles, the number of mature eggs collected, the quality of developing embryos, and early pregnancy outcomes. No additional procedures or medications will be required beyond standard IVF care. The goal is to better understand whether adding recombinant LH provides any measurable benefit in dydrogesterone-based PPOS cycles.

DETAILED DESCRIPTION:
This prospective observational study aims to evaluate how two routinely used gonadotropin strategies influence ovarian response and reproductive outcomes in women undergoing IVF treatment with a dydrogesterone-based Progestin-Primed Ovarian Stimulation (PPOS) protocol. In standard clinical practice, ovarian stimulation may be performed using recombinant FSH alone or a combination of recombinant FSH and recombinant LH. Both approaches are already used in daily care, and the choice of regimen is determined by the treating physician according to individual patient characteristics. The study does not assign treatments; instead, it observes and compares outcomes in patients receiving these medications as part of routine management.

Dydrogesterone is administered from Day 2 of the cycle to prevent premature LH surges, allowing controlled follicular growth. Participants will undergo regular ultrasound monitoring and bloodwork as part of their usual IVF treatment. When appropriate follicular maturation is achieved, final oocyte maturation will be triggered, followed by oocyte retrieval according to standard clinical protocols.

The primary focus of this study is to compare the number of mature (MII) oocytes obtained between the two gonadotropin regimens. Secondary outcomes include the number of good-quality blastocysts, implantation rate, and ongoing pregnancy rate, which together provide a comprehensive assessment of IVF success. Additional stimulation characteristics-such as follicle growth patterns, estradiol and LH levels, total gonadotropin dose, and duration of stimulation-will also be documented to explore differences in cycle dynamics.

No extra medications, procedures, or interventions will be required beyond routine IVF care. All data will be collected prospectively and analyzed to determine whether adding recombinant LH offers measurable clinical advantages compared with recombinant FSH alone in dydrogesterone-PPOS cycles.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20 to 43 years.
* BMI < 30 kg/m².
* AMH > 1 ng/mL.
* Undergoing IVF/ICSI treatment with a dydrogesterone-based PPOS protocol.
* Women with regular menstrual cycles or clinically acceptable cycle pattern for stimulation.
* Ability to provide informed consent and comply with study procedures.
* Presence of at least one ovary and eligibility for controlled ovarian stimulation

Exclusion Criteria:

* Cycle cancellation due to lack of viable embryos.
* Prior or planned PGT-A in the same cycle.
* Adenomyosis diagnosed by ultrasound or MRI.
* Uncorrected uterine anomalies (e.g., bicornuate, unicornuate, didelphys uterus).
* Presence of hydrosalpinx.
* Use of oral contraceptives or luteal-phase estradiol within 3 months before stimulation.
* Refusal or inability to provide informed consent.
* Severe systemic disease or contraindication to ovarian stimulation.
* Prior bilateral oophorectomy

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be selected from women seeking infertility treatment at a fertility clinic and undergoing in-vitro fertilization (IVF) with controlled ovarian stimulation. This population typically consists of reproductive-age women who have difficulty achieving pregnancy and require assisted reproductive technologies. Eligible patients are generally healthy enough to undergo ovarian stimulation, have adequate ovarian reserve (AMH > 1 ng/mL), and meet age and BMI criteria for standard IVF care. Women in this group routinely receive dydrogesterone-based PPOS protocols as part of their clinical treatment, and the choice of gonadotropin regimen (rFSH alone or rFSH+rLH) follows routine medical practice. This population reflects real-world patients commonly treated in IVF programs
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
mature oocytes collected (MII) | The overall assessment period spans the duration of ovarian stimulation and scheduling of oocyte aspiration, with a maximum observation period of up to 3-4 weeks
  Time Frame:
  From the date of participant enrollment, including initiation of controlled ovarian stimulation, through the completion of the oocyte pick-up (OPU) procedure, with the number of mature (metaphase II) oocytes assessed and recorded exclusively at the time of oocyte aspiration. The overall assessment period spans the duration of ovarian stimulation and scheduling of OPU, with a maximum observation period of up to 3-4 weeks

SECONDARY OUTCOMES:
total numbers of blastocysts | From participant enrollment and initiation of ovarian stimulation through completion of embryo culture to the blastocyst stage, over a maximum period of up to 3-4 weeks.
  The total number of blastocyst-stage embryos generated per cycle, defined as embryos that reach the blastocyst stage (Day 5 or Day 6) following in vitro fertilization or intracytoplasmic sperm injection (ICSI), and recorded after completion of embryo culture.
  Time Frame
  From the date of participant enrollment, including initiation of controlled ovarian stimulation, through completion of embryo culture to the blastocyst stage, with the total number of blastocysts assessed and recorded after final blastocyst evaluation (Day 5-6 embryo culture). The overall assessment period includes ovarian stimulation, oocyte pick-up (OPU), fertilization, and extended embryo culture, with a maximum observation period of up to 3-4 weeks.
numbers of top quality blastocysts | Day 5 after fertilization
  Top-quality blastocysts are defined according to the Gardner and Schoolcraft blastocyst grading system as blastocysts with full expansion (grade ≥3), an inner cell mass (ICM) grade of A or B, and a trophectoderm (TE) grade of A or B (i.e., grades ≥3BB)
Clinical pregnancy rate per embryo transfer | 6-7 weeks after embryo transfer
  Clinical pregnancy rate per embryo transfer is defined as the proportion of embryo transfer cycles resulting in at least one intrauterine gestational sac with fetal cardiac activity confirmed by transvaginal ultrasound.
  Unit: %
Live birth rate per embryo transfer (LBR per ET) | At delivery
  Live birth rate per embryo transfer is defined as the proportion of embryo transfer cycles resulting in the delivery of at least one live-born infant after ≥24 weeks of gestation.
  Unit: percentage

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Centrum Clinic IVF Center, Ankara, Ankara
  - Bahçeci IVF Center, Ankara

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves sensitive reproductive health information and data are collected solely for clinical and research purposes within the center. Only aggregated, de-identified results will be reported in publications.
  Supporting Documents to Be Shared: None.

REFERENCES:
- [Background] Muharam R, Nurdya AN, Yo EC, Sumapraja K, Harzif AK, Maidarti M, Wiweko B, Hestiantoro A. Comparing Dydrogesterone Versus Medroxyprogesterone in Progestin-Primed Ovarian Stimulation (PPOS) for Patients Undergoing In Vitro Fertilization/Intracytoplasmic Sperm Injection: A Systematic Review. Cureus. 2025 Jun 13;17(6):e85959. doi: 10.7759/cureus.85959. eCollection 2025 Jun. PMID 40524846
- [Background] Zhang J, Du M, Li Z, Liu W, Ren B, Zhang Y, Guan Y. Comparison of Dydrogesterone and Medroxyprogesterone in the Progestin-Primed Ovarian Stimulation Protocol for Patients With Poor Ovarian Response. Front Endocrinol (Lausanne). 2021 Sep 24;12:708704. doi: 10.3389/fendo.2021.708704. eCollection 2021. PMID 34630325
- [Background] Yu S, Long H, Chang HY, Liu Y, Gao H, Zhu J, Quan X, Lyu Q, Kuang Y, Ai A. New application of dydrogesterone as a part of a progestin-primed ovarian stimulation protocol for IVF: a randomized controlled trial including 516 first IVF/ICSI cycles. Hum Reprod. 2018 Feb 1;33(2):229-237. doi: 10.1093/humrep/dex367. PMID 29300975